CLINICAL TRIAL: NCT03740620
Title: The Effect of Bevel Direction on the Pathway of the Tracheal Tube in the Nasal Cavity During Nasotracheal Intubation: a Randomized Controlled Trial
Brief Title: The Effect of Bevel Direction on the Pathway of the Nasotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 30-2018-76
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Epistaxis; Intubation Complication
Keywords: epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): In the intervention group, a nasotracheal tube is inserted into the nostril with the bevel of the tube facing the cephalad direction of the patient.
  Interventions: Procedure: Bevel facing the cephalad direction of the patient
- conventional group (Active Comparator): In the conventional group, a nasotracheal tube is inserted in a usual way, i.e., with the bevel of the tube facing the left side of the patient.
  Interventions: Procedure: Bevel facing leftward of the patient

INTERVENTIONS:
Procedure: Bevel facing the cephalad direction of the patient — The bevel of the nasotracheal tube facing cephalad direction of the patient
  Arms: intervention group
Procedure: Bevel facing leftward of the patient — The bevel of the nasotracheal tube facing the left side of the patient
  Arms: conventional group

SUMMARY:
In this study, the subjects are divided into two groups (group I: intervention group = the nasotracheal tube inserted with the bevel of the nasal tube facing the direction of the patient's head, and Group II: conventional group = the bevel of the tube toward the left side of the subject). After the endotracheal tube is introduced, a flexible endoscope is used to evaluate whether the tube is located below the inferior turbinate, i.e. in the lower pathway.

DETAILED DESCRIPTION:
Primary outcome

* incidence of tracheal tube passing through the lower pathway (beneath the inferior turbinate and immediately above the nasal floor of the nostril) Secondary outcome
* intubation time
* incidence of epistaxis
* severity of bleeding
* Resistance during Insertion of the tracheal tube

ELIGIBILITY:
Inclusion Criteria:

* a patient who will take operation which needs nasotracheal intubation under general anesthesia

Exclusion Criteria:

* a patient who didn't agree to participate in this study
* a patient who has a deformity of the nose
* a patient who has a history of severe epistaxis
* a patient who has coagulation problem
* a patient who has a history of the fracture or surgery of the skull base

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
incidence of the tube in lower pathway | right after completion of the intubation
  incidence of tracheal tube passing through the lower pathway (beneath the inferior turbinate and immediately above the nasal floor of the nostril)

SECONDARY OUTCOMES:
intubation time | from the start of the intubation to the completion of the intubation, which is confirmed by the appearance of end-tidal CO2 curve, up to 60 seconds
  time to complete endotracheal intubation
incidence and severity of epistaxis | right after completion of the intubation
  incidence and severity of epistaxis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Won D, Kim H, Chang JE, Lee JM, Min SW, Jung J, Yang HJ, Hwang JY, Kim TK. Effect of bevel direction on the tracheal tube pathway during nasotracheal intubation: A randomised trial. Eur J Anaesthesiol. 2021 Feb 1;38(2):157-163. doi: 10.1097/EJA.0000000000001347. PMID 33009189